CLINICAL TRIAL: NCT04957459
Title: Prospective, Observational,Non-interventional Research of The Correlation of Preoperative Measurement Parameter on the Predicting of Visual Outcomes Among Patients With Idiopathic Macular Holes
Brief Title: The Correlation of Preoperative Measurement Parameter on the Predicting of Visual Outcomes Among Patients With Idiopathic Macular Holes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: I2021001380
Record Dates: First submitted 2021-06-08; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Macular Holes
Keywords: idiopathic full thickness macular hole; OCTA; postoperative best corrected visual acuity; vitrectomy
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study retrospectively analyzed the relationship between the preoperative optical coherence tomography(OCT) and optical coherence tomography angiography(OCTA) software related parameters of patients with idiopathic macular hole, the patient's own clinical data and the best corrected visual acuity (BCVA) for at least one month after surgery.

DETAILED DESCRIPTION:
After Pars plana vitrectomy combined with removal of the internal limiting membrane (ILM) and air filling, it can not only promote the closure of the macular hole in patients with idiopathic macular hole, but also improve the visual acuity of the affected eye. There are various studies to predict the visual acuity of patients after surgery recovery, but due to many factors that affect the effect of macular hole surgery, the improvement of visual acuity after retinal surgery varies greatly in different eyes. As a new type of ophthalmology device, OCTA plays an important role in measuring the size of the hole and the changes of retinal capillaries. Therefore, this study intends to calculate patient parameters based on OCT and OCTA equipment. Statistical software was used to analyze the relationship between each parameter and the best corrected visual acuity (BCVA) for at least one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic MHs, the MH is closed ,and follow-up for at least 1 month after vitrectomy.

Exclusion Criteria:

* High myopia (≥6 diopters,AL≥26.5mm), increased intraocular pressure (IOP, >21 mm Hg) or glaucoma, severe cataract, severe corneal disease，severe systemic conditions that prevent surgery, and history of ocular trauma, intraocular inflammation, retinal vascular disease, or previous ocular surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic macular hole after vitrectomy combined with internal limiting membrane peeling and air-filling surgery and the MH is closed and the postoperative best corrected visual acuity is at least 1 month
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Macular hole status | at 1 month after surgery
  macular hole status (open, flat open or closed)
MLD of macular hole | Before surgery
  Calculation of minimum liner diameter of macular hole with optical coherence tomography angiography
BD of macular hole | Before surgery
  Calculation of base diameter of macular hole with optical coherence tomography angiography
Choroidal hypertransmission width of macular hole | Before surgery
  Calculation of Choroidal hypertransmission width of macular hole with optical coherence tomography angiography
Horizontal ellipsoid band missing diameter of macular hole | Before surgery
  Calculation of Horizontal ellipsoid band missing diameter of macular hole with optical coherence tomography angiography
Baseline best-corrected visual acuity | Before surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
best-corrected visual acuity at 1 month | at 1 month after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
best-corrected visual acuity at 2 months | at 2 months after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
best-corrected visual acuity at 3 months | at 3 months after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
best-corrected visual acuity at 4 months | at 4 months after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
best-corrected visual acuity at 5 months | at 5 months after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
best-corrected visual acuity at 6 months | at 6 months after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
FAZ area of macular hole | Before surgery
  Calculation of foveal avascular zone (FAZ) area of macular hole with optical coherence tomography angiography
FAZ area of macular hole at 1 month | at 1 month after surgery
  Calculation of foveal avascular zone (FAZ) area of macular hole with optical coherence tomography angiography
FAZ area of macular hole at 2 months | at 2 months after surgery
  Calculation of foveal avascular zone (FAZ) area of macular hole with optical coherence tomography angiography
FAZ area of macular hole at 3 months | at 3 months after surgery
  Calculation of foveal avascular zone (FAZ) area of macular hole with optical coherence tomography angiography
FAZ area of macular hole at 4 months | at 4 months after surgery
  Calculation of foveal avascular zone (FAZ) area of macular hole with optical coherence tomography angiography
FAZ area of macular hole at 5 months | at 5 months after surgery
  Calculation of foveal avascular zone (FAZ) area of macular hole with optical coherence tomography angiography
FAZ area of macular hole at 6 months | at 6 months after surgery
  Calculation of foveal avascular zone (FAZ) area of macular hole with optical coherence tomography angiography
CRT of macular hole | Before surgery
  Calculation of central retinal thickness(CRT) of macular hole with optical coherence tomography angiography
CRT of macular hole at 1 month | at 1 month after surgery
  Calculation of central retinal thickness(CRT) of macular hole with optical coherence tomography angiography
CRT of macular hole at 2 months | at 2 months after surgery
  Calculation of central retinal thickness(CRT) of macular hole with optical coherence tomography angiography
CRT of macular hole at 3 months | at 3 months after surgery
  Calculation of central retinal thickness(CRT) of macular hole with optical coherence tomography angiography
CRT of macular hole at 4 months | at 4 months after surgery
  Calculation of central retinal thickness(CRT) of macular hole with optical coherence tomography angiography
CRT of macular hole at 5 months | at 5 months after surgery
  Calculation of central retinal thickness(CRT) of macular hole with optical coherence tomography angiography
CRT of macular hole at 6 months | at 6 months after surgery
  Calculation of central retinal thickness(CRT) of macular hole with optical coherence tomography angiography

CONTACTS AND LOCATIONS:
Overall Officials: Qi Wan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Department of Ophthalmology, The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No